CLINICAL TRIAL: NCT05817825
Title: Pilot Testing a Novel Remotely Delivered Intensive Outpatient Program for Individuals With Opioid Use Disorder Hospitalized With Serious Injection-related Infection
Brief Title: Pilot Testing a Novel Remotely Delivered Intensive Outpatient Program for Individuals With OUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Mclean Hospital (Other)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Director, Division of Addiction Psychiatry, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P000709; R21DA056799 (NIH)
Record Dates: First submitted 2023-03-07; First posted 2023-04-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Opioid Use Disorder; Serious Bacterial Infections
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: The trial is an open-label, single-arm, pilot feasibility trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): The intervention to be developed and tested has two components: 1) the remotely delivered IOP ("Smart IOP"), and 2) a peer recovery coach to provide support and accountability to the participant.
  Interventions: Behavioral: Smart IOP Intervention; Behavioral: Peer Recovery Coach

INTERVENTIONS:
Behavioral: Smart IOP Intervention — Smart IOP is a remotely delivered IOP program in operation since 2016, allowing patients to complete addiction treatment entirely online. The original program, consisting of 72 video modules across 8 different topics, will be adapted and tailored to hospitalized patients with serious infections from injection drug use. Participants will watch video content asynchronously, and will be required to correctly answer knowledge questions to proceed to the next module. The whole treatment program will require approximately 4 weeks to complete. Participants are also asked to answer questions about how to apply the knowledge to their own personal circumstances. The answers to these are reviewed by the peer recovery coach during weekly encounters. Videos can be viewed at a time that is most convenient to the participants. T
Behavioral: Peer Recovery Coach — Peer recovery coach, an individual in sustained recovery (>5 years) and certified to be a coach, will meet weekly with the participant to review progress, answer questions about the videos, review answers to questions, and encourage continuation of treatment after discharge. These meetings will occur in-person or remotely.

SUMMARY:
This study aims to test a remotely delivered IOP program ("SmartIOP") for OUD patients who are hospitalized for serious injection-related infections. This will be a pilot trial to assess the feasibility of the IOP program and examine OUD-related outcomes following discharge from the hospital.

DETAILED DESCRIPTION:
The aim is to conduct a single-arm pilot study of 20 participants who are hospitalized for serious injection-related infections to complete the newly tailored program. The intervention to be developed and tested has two components: 1) the remotely delivered IOP ("Smart IOP"), and 2) a peer recovery coach who will provide support and accountability to the participant. The feasibility of the intervention will be established by evaluating recruitment and the acceptability of the program according to a priori benchmarks. The study team will assess the program's preliminary efficacy by evaluating OUD-related outcomes for up to 28 days after discharge from the hospital. The study will be conducted at Brigham and Women's Hospital (BWH), an urban, 793-bed academic medical center located in Boston, MA, and a major teaching hospital for Harvard Medical School.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults aged 18 and above
* Any DSM-5 substance use disorder
* Can identify at least 2 individuals who can act as points of contact following discharge from the hospital

Exclusion Criteria:

* Psychotic disorder, active suicidality, or homicidally
* Condition likely to be terminal during the study period
* Unable to perform consent due to impaired mental status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention program | Immediately Post Intervention
  We expect the results to demonstrate adequate feasibility, as defined by exceeding the threshold for adequate recruitment feasibility and good program acceptability. Adequate recruitment feasibility is defined as enrolling more than 70% of those eligible individuals. Excellent program acceptability is defined as >70% of the participants complete at least 70% of the Smart IOP intervention, and good program acceptability if >60% of participants did.

SECONDARY OUTCOMES:
Illicit opioid use | 7-day Follow Up, 14-day Follow Up, 21-day Follow Up, and 28-Day Follow Up
  As an exploratory outcome, we will evaluate, using the Timeline follow back (TLFB), the proportion of days using illicit opioids during the follow-up period compared to baseline.
Retention with MOUD treatment | 7-day Follow Up, 14-day Follow Up, 21-day Follow Up, and 28-Day Follow Up
  As an exploratory outcome, we will evaluate the proportion of participants who successfully engaged with addiction treatment following completion of the intervention compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States